CLINICAL TRIAL: NCT07213037
Title: Magnesium Sulfate Versus Lidocaine as Additives to Dexmedetomidine for Cough Suppression After Functional Endoscopic Sinus Surgery
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Aboelmaged Abdelmawjoud, residant doctor at Assiut university hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Magnesium Sulfate vs Lidocaine
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Cough Suppression
MeSH Terms: interventions — Dexmedetomidine; Magnesium Sulfate; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Active Comparator): patients will be given intravenous dexmedetomidine plus magnesium sulphate
  Interventions: Drug: Dexmedetomidine; Drug: Magnesium sulfate
- Group B (Active Comparator): patients will be given intravenous dexmedetomidine plus lidocaine
  Interventions: Drug: Dexmedetomidine; Drug: lidocaine

INTERVENTIONS:
Drug: Dexmedetomidine — patients will receive dexmedetomidine(D) in dose 0.2 μg/kg/h infusion via syringe pump during surgery
Drug: Magnesium sulfate — patients will be given intravenous dose 30mg/kg.
  Arms: Group A
Drug: lidocaine — patients will be given in one dose 1.5 mg/kg.
  Arms: Group B

SUMMARY:
Functional Endoscopic Sinus Surgery (FESS) is a widely performed procedure for the management of chronic rhinosinusitis and nasal polyposis. Despite being minimally invasive(1).Postoperative coughing, in particular, is a frequent complication that can increase venous pressure, disrupt the surgical site, cause bleeding, and prolong recovery(2).

Coughing and other airway reflexes during extubation are largely mediated by the stimulation of rapidly adapting stretch receptors (RARs) in the trachea, often aggravated by the presence of an endotracheal tube(3). Although these reflexes are suppressed under deep anesthesia, they become prominent as the patient regains consciousness. A smooth and controlled emergence from anesthesia is especially important in sinonasal procedures where postoperative bleeding can have serious consequences(4).

Postoperative sore throat (POST) is considered a minor complication of general anesthesia. POST complaints can range in severity from slight throat irritation to incapacitating discomfort that prevents swallowing, and transitory voice alterations are frequently noticed during the postoperative visit. The identified risk factors for POST following tracheal intubation include female gender, younger age, preexisting lung disease, longer anesthesia duration, and blood-stained endotracheal tube (ETT) at extubation. The ETT size, intubation techniques, and muscle relaxant use are also associated with POST development(5).

Dexmedetomidine, a highly selective alpha-2 adrenergic agonist, has emerged as another promising agent for attenuating airway reflexes. It provides sedative, anxiolytic, and sympatholytic effects without significant respiratory depression(6). Dexmedetomidine reduces central sympathetic output and modulates the arousal pathways, leading to smoother emergence and decreased airway hyperreactivity. Its ability to suppress extubation-related coughing has been demonstrated in several clinical studies, along with favorable effects on hemodynamic stability and postoperative analgesia(7).

Among the strategies employed to reduce this airway reactivity is intravenous (IV) lidocaine, it has been used effectively to blunt airway reflexes(8). It exerts its action by stabilizing neuronal membranes and inhibiting sodium channel activity, thereby decreasing the excitability of afferent airway nerves(9). IV lidocaine also reduces mucus secretion and limits tracheal irritation, resulting in fewer instances of coughing and sore throat. Its safety profile, rapid onset, and ease of administration make it a practical choice in a variety of surgical settings.

Magnesium sulfate, which acts as an NMDA receptor antagonist, is currently recognized as one of the most effective agents for the prevention and management of POST by peripheral NMDA receptors. Local application of magnesium can mitigate nociceptive stimuli caused by mucosal inflammation triggered by endotracheal intubation. Magnesium sulfate also exhibits, anti-inflammatory, and anti-edema properties for traumatic edema and inflammation(10).

Despite the individual benefits of lidocaine, Magnesium sulfate and dexmedetomidine, there is limited direct comparative data regarding their relative efficacy in preventing postoperative cough following FESS.

ELIGIBILITY:
Inclusion Criteria:

* a. Age >18 < 60 years old b. Both genders. c. Patients who were in risk-scoring groups I-II of the American Society of Anesthesiologists (ASA)

Exclusion Criteria:

* . Active airway infection
* History of tracheal and laryngeal surgery.
* Airway tumors,
* Body mass index more than 35.
* Increased intracranial and intraocular pressure.
* Uncontrolled pulmonary diseases (bronchial asthma, chronic obstructive pulmonary disease (COPD), restrictive lung diseases).
* Patients with a known allergy or sensitivity to any study drugs.
* Patients' refusal to enroll in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
severity of postoperative cough | 24 hours
  severity of cough was graded as follows: grade 0 = no cough; grade 1 =single cough; grade 2 = more than one attack of non-sustained cough; grade 3 = repeated and sustained cough with head lift